CLINICAL TRIAL: NCT02874638
Title: Effect of Non-essential Amino Acids on Protein Requirements for Endurance Athletes Using Indicator Amino Acid Oxidation Method.
Brief Title: Effect of Non-essential Amino Acids on Protein Requirements for Endurance Athletes
Acronym: EA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IAAO-EA3
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- BASE egg protein (Experimental): 0.8 g/kg/d of BASE protein provided as crystalline amino acid made after egg protein.
  Interventions: Dietary Supplement: BASE egg protein
- BCAA-enriched egg protein (Experimental): branched-chain amino acid-enriched egg protein
  Interventions: Dietary Supplement: BCAA-enriched egg protein
- small amount of essential amino acids (Experimental): small amount of essential amino acids made after egg protein, which is equivalent to the amount of essential amino acids in BASE
  Interventions: Dietary Supplement: small amount of essential amino acids
- large amount of essential amino acids (Experimental): large amount of essential amino acids made after egg protein, which is equivalent to the amount of amino acids in BCAA
  Interventions: Dietary Supplement: large amount of essential amino acids

INTERVENTIONS:
Dietary Supplement: BASE egg protein — 0.8 g/kg/d of protein provided as crystalline amino acid modeled after egg protein
  Arms: BASE egg protein
Dietary Supplement: BCAA-enriched egg protein — BCAA-enriched egg protein provided as crystalline amino acid.
  Arms: BCAA-enriched egg protein
Dietary Supplement: small amount of essential amino acids — essential amino acids modeled after egg protein, provided as crystalline amino acid, which is equivalent to the amount of essential amino acid in BASE egg protein
  Arms: small amount of essential amino acids
Dietary Supplement: large amount of essential amino acids — essential amino acids modeled after egg protein, provided as crystalline amino acid, which is equivalent to the amount of amino acid in BCAA-enriched egg protein
  Arms: large amount of essential amino acids

SUMMARY:
Protein requirements in individuals who participate in endurance-based exercise training have been suggested to be greater than the current recommended dietary allowance (RDA).

The biological value of protein depends on its amino acid composition. Essential amino acids are believed to have main role on whole body protein metabolism. However, it remains to be determined what role non-essential amino acids (NEAA) may have in regulating protein metabolism and contributing to the increased protein requirements after endurance exercise.

The indicator amino acid oxidation (IAAO) method has clarified the individual amino acid requirement in children, normal healthy adult and clinical populations. However, the IAAO method has never been utilized for assessing the effect of NEAA on protein requirements after endurance exercise.

The objective of the current study is to investigate the importance of NEAA for endurance-trained male subjects.

ELIGIBILITY:
Inclusion Criteria:

* endurance-trained participants who regularly run more than 40 km/week
* Participants who are categorized at least "very good" based on a study by Shvartz & Reibold, in which VO2peak is used as an index. (i.e. the participants whose VO2peak is ≥57 ml/kg/min (18-24 y), ≥54 ml/kg/min (25-29 y), ≥52 ml/kg/min (30-34 y), ≥49 ml/kg/min (35-39 y)
* Ability to complete the 16-km familiarization run in session 2

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the physical activity readiness questionnaire (PAR-Q+)
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
13CO2 (carbon dioxide) excretion rate (μmol/kg/h) | at 8 hours after the end of exercise]
  8 hours after exercise followed by ingesting 13C-labelled phenylalanine and one of 5 different amount of amino acids intake, 13CO2 excretion rate is determined by multiplying the enrichment of 13CO2 in breath measured by Mass spectrometry and CO2 production rate measured by metabolic cart.

SECONDARY OUTCOMES:
[13C]phenylalanine oxidation rate (μmol/kg/h) | at 8 hours after the end of exercise
  8 hours after exercise followed by ingesting 13C-labelled phenylalanine and one of 5 different amount of amino acids intake, 13CO2 excretion rate is determined dividing 13CO2 excretion rate by urinary enrichment of 13C-phenylalanine in breath measured by Mass spectrometry, and CO2 production rate measured by metabolic cart.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Ph.D., Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No